CLINICAL TRIAL: NCT03705299
Title: A Prospective, Comparative Study to Evaluate the Accuracy of a Non-Invasive Central Venous Pressure Method to the Standard CVP Method
Brief Title: Non-Invasive CVP Method to Standard CVP Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: NeuroDx Development (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-121
Record Dates: First submitted 2018-06-19; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-07

CONDITIONS: Central Venous Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NeuMeDex NICVP (Non-Invasive CVP) vs Standard CVP (Experimental): Three pressure readings recorded for both NeuMeDex NICVP and central line pressure catheter over a 10 minute period.
  Interventions: Device: Non-Invasive CVP vs Standard CVP

INTERVENTIONS:
Device: Non-Invasive CVP vs Standard CVP

SUMMARY:
This is a prospective, comparative, internally controlled device study that will enroll a total of 100 adult patients that require the placement of central venous catheter and CVP monitoring to assess volume status and cardiac preload.

DETAILED DESCRIPTION:
Standard CVP Method

The CVP line is inserted into the internal jugular vein central venous catheter or subclavian vein catheter and threaded to the point where the superior vena cava meets the inferior vena cava prior to entry into the right atrium of the heart. The catheter is hooked to a pressure bag which is pressurized to 200 cm water. This pressure allows the infusion of about 3ml of fluid each hour but keeps the line patent. The distal tip of the CVP line is connected to a transducer and taped to the arm at a level which is in line with the heart.

Research Procedure (non-invasive CVP Method)

A physiologic data acquisition system (Zoe Medical, Topsfield MA)) will be used to monitor CVP, upper arm impedance changes, and upper arm cuff pressures.

The subject's CVP pressure transducer will be zeroed at the level of the right atrium (midaxillary line) with the use of a carpenter's level.

A tetra-polar impedance configuration will be used to measure upper arm impedance. A pair of current-injecting electrodes will be placed in positions 1 & 4 and two sensing electrodes will be placed in positions 2 & 3 (where a traditional blood pressure cuff would be positioned, overlying the brachial-axillary vein system). These leads extend from the Zoe Medical device. (Figure 1 taken from Ward et al., in press).

Electrobioimpedance will be measured in the upper portion of an upper extremity using an electrobioimpedance amplifier contained within the Zoe Medical device. A constant current source (1mA, 100kHz) will be sent through the current electrode and the voltage drop between the two sensing electrodes will be amplified.

A blood pressure cuff attached to the Zoe Medical Device will be positioned over the two sensing electrodes.

The cuff pressure will be quickly inflated to a value higher than CVP but lower than the diastolic arterial pressure (40 mm Hg) and kept at that pressure for 45-60 seconds.

At the end of the inflation hold period, release the cuff pressure valve and open to atmosphere to allow rapid self-deflation

Repeat measures 3 times in each subject for a period of 10 minutes

If the subject requires volume resuscitation, diuresis, or are administered inotropic drugs, we will reevaluate CVP with the non-invasive method during these circumstances. CVP will be measured every 1 minute to capture rapid changes in CVP. The length of time that the investigators monitor CVP will depend on the length of time required to detect changes in CVP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Require CVP monitoring in the supine position as part of routine care
* Central venous access obtained by either internal or external jugular, or subclavian vein

Exclusion Criteria:

* Patients aged < 18 years
* Patients who are pregnant
* Patients that will be in the prone position
* Central venous access obtained by the femoral vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Assessing if the NeuMeDx NICVP device is as effective as the standard invasive method at measuring CVP in patients that require central catheter placement and monitoring. | 6 months
  The primary objective of the study is to measure the CVP using the NeuMeDx NICVP (Non-Invasive Central Venous Pressure) device. The critical endpoint is the average of the average of three CVP, by calibrated forced transducer, and NICVP measurements in mmHg over a 10-minute period in a patient in the supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Gratz, DO, Principal Investigator — The Cooper Health System

IPD SHARING:
Plan to Share IPD: No